CLINICAL TRIAL: NCT05325359
Title: Validity and Reliability of L Test in Persons With Multiple Sclerosis
Brief Title: L Test in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Furkan BİLEK, Lecturer, Firat University
Other Study IDs: Fırat Univers
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Balance; L test; Validity; Gait
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple sclerosis: . Inclusion criteria for volunteers; Individuals with relapsing-remitting type MS, who are between 18-65, EDSS scores between 1 ≤ and ≤ 5.5, individuals who score 24 and above in Mini Mental State Examination and who can walk a minimum of 20 m independently will be included. In addition, exclusion criteria for volunteers; Severe spasticity of the lower extremities (Ashworth score 3 or 4), having an acute MS attack or a history of an attack in the last 1 month, having an orthopedic or systemic problem that would prevent participation in the tests, having another neuromuscular disorder other than MS, visual involvement or diplopia, and is that he has a cardio-pulmonary problem that will prevent him from participating in the tests.
  Interventions: Behavioral: L test

INTERVENTIONS:
Behavioral: L test — It is an expanded version of the TUG and is designed to assess advanced functional ambulation with more detail available elsewhere. It is recorded when the participant gets up from the chair, walks 3 m to a cone, turns 90° to the right, continues to walk 7 m to the next cone, turns 180° left around the cone, then returns to the chair the same way. The test time is recorded, starting with the word "go" and ending with the participant's back touching the back of the chair.

SUMMARY:
Multiple Sclerosis (MS), a chronic inflammatory disease of the central nervous system, is a disease characterized by myelin, oligodendrocyte and axon damage [1]. Research continues on the autoimmune, infectious, environmental, vascular and genetic origins of this disease, which affects approximately 2.5 million people in the world and is seen 2-3 times more in women than in men. Although the signs and symptoms of the disease vary according to the location of the lesion; Loss of balance and strength, spasticity, sensory disturbances, fatigue, ataxia, autonomic dysfunction, and decreased visual acuity is frequently observed.

There are no studies in the literature investigating the validity and reliability of this test in individuals with MS. Reliability is population-specific and it is important to investigate the reliability of the L test in MS patients. Therefore, the aim of our study is to reveal the test-retest reliability and validity of the L test.

DETAILED DESCRIPTION:
General Information about the Research, Rationale and Objectives:

Multiple Sclerosis (MS), a chronic inflammatory disease of the central nervous system, is a disease characterized by myelin, oligodendrocyte and axon damage [1]. Research continues on the autoimmune, infectious, environmental, vascular and genetic origins of this disease, which affects approximately 2.5 million people in the world and is seen 2-3 times more in women than in men [1, 2]. Although the signs and symptoms of the disease vary according to the location of the lesion; Loss of balance and strength, spasticity, sensory disturbances, fatigue, ataxia, autonomic dysfunction, and decreased visual acuity are frequently observed [1].

Abnormalities and losses in balance management are frequently seen in individuals with MS [3-6] . This abnormality, together with other risk factors, increases the risk of falling [7] and causes limitations in patients' activities of daily living. Studies on balance problems in elderly individuals are frequently investigated in the literature. However, the frequency of falls in this population was found to be 1.5 falls per year [8], while another study investigating individuals with MS found an average of 9 falls per year [7]. In order to develop fall prevention or reduction strategies, it is necessary to evaluate different aspects of motor impairment and to accurately identify factors contributing to falls [9-11]. Since falls among MS patients have a multifactorial etiology, multiple evaluations are necessary to explore the balance problem.

Although various scales have been developed to evaluate the functional level of MS patients [12, 13], the use of frequently applied scales in this patient group allows the results to be compared with other studies and other pathologies. In addition, the use of frequently applied scales does not require special training of raters. Previous studies have used the Berg Balance Scale, the Functional Reach Test, the Timed Get Up and Walk test, and general measures of fall risk (eg, questioning the date of fall) [14-16]. These tests primarily assess the ability to walk forward, turn back, and take a step.

The reliability of the TUG in people with MS has ranged from 'good' to 'excellent' [17,18], but the TUG is only an opportunity for unilateral disorders to turn in a preferred direction [19]. Thus, despite good reliability and validity, TUG currently has limitations in MS that can only be overcome by adding complex and potentially excessively expensive instrumentation. The L test is a modification of the TUG that extends the walking distance from 6 to 20 m and also requires participants to make both clockwise and counterclockwise turns. Therefore, it may have limited sensitivity and the potential to overcome ceiling effects. The L test was originally designed for individuals following lower limb amputation and has since been evaluated in stroke and hospitalized elderly subjects [19-21]. In all three studies, the L test showed good reliability and also showed good correlation with the TUG. The aim of this study is to evaluate the L test in terms of test/retest reliability and concurrent validity with TUG in individuals with MS. There are no studies in the literature investigating the validity and reliability of this test in individuals with MS. Reliability is population specific and it is important to investigate the reliability of the L test in MS patients. Therefore, the aim of our study is to reveal the test-retest reliability and validity of the L test.

10. Detailed Material and Methodology of the Research: The methodological model of the study is the validity and reliability study. Our study will include individuals who applied to Fırat University Training and Research Hospital after ethical approval and were diagnosed with Relapsin-Remitting MS by a neurologist. It is planned to collect the Helsinki Declaration on a voluntary basis from individuals whose data meet the inclusion criteria. As demographic characteristics; The age, gender, body weight, height, EDSS score, occupation and education level of the patients, the history of the disease, the number of falls in the last year and the type of MS will be recorded. Inclusion criteria for volunteers; Individuals with relapsing-remitting type MS, who are between 18-65, EDSS scores between 1 ≤ and ≤ 5.5, individuals who score 24 and above in Mini Mental State Examination and who can walk a minimum of 20 m independently will be included. In addition, exclusion criteria for volunteers; Severe spasticity of the lower extremities (Ashworth score 3 or 4), having an acute MS attack or a history of an attack in the last 1 month, having an orthopedic or systemic problem that would prevent participation in the tests, having another neuromuscular disorder other than MS, visual involvement or diplopia, and is that he has a cardio-pulmonary problem that will prevent him from participating in the tests.

Our study will be carried out as a "test-retest" design and the psychometric properties of the L test in MS patients will be examined. 3 m walk back test, Timed Up and Go, 4-Square Step Test test will be applied to the patients. All assessments will be done by the same physiotherapist. The second evaluation will be performed by the same physiotherapist two days after the first evaluation (test) to measure test-retest reliability. Data collection with the same rater will be preferred to avoid inter-rater variability and error rate between evaluations.

According to Lexell and Downham, 30-50 participants should be included in reliability studies [22]. Considering this recommendation, which defines the reliability of the L test, it is planned to include 50 individuals with MS in our study.

L Test; It is an expanded version of the TUG and is designed to assess advanced functional ambulation with more detail available elsewhere. It is recorded when the participant gets up from the chair, walks 3 m to a cone, turns 90° to the right, continues to walk 7 m to the next cone, turns 180° left around the cone, then returns to the chair the same way. The test duration is recorded, beginning with the word "go" and ending with the participant's back touching the back of the chair [23].

3-meter Walk Back Test; The 3-meter distance is marked with a black tape and participants are asked to align their heels with the black tape. Individuals are asked to walk backwards as soon as possible with the "walk" command and stop when they reach 3 meters. Meanwhile, the elapsed time is recorded in seconds. Evaluation will be done three times and the average time will be recorded [24].

Timed Get Up and Go Test; It is applied to assess the balance and fall risk of individuals. The patient is first asked to sit leaning on the chair. The patient is then asked to stand up, walk with regular steps for a predetermined distance of 3 meters, return at the end of 3 meters and sit in a chair. During the test, the patient's walking time is recorded in seconds with a stopwatch. The test was repeated three times and the mean value will be recorded [25].

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for volunteers; Individuals with relapsing-remitting type MS, who are between 18-65, EDSS scores between 1 ≤ and ≤ 5.5, individuals who score 24 and above in Mini Mental State Examination and who can walk a minimum of 20 m independently will be included.

Exclusion Criteria:

* In addition, exclusion criteria for volunteers; Severe spasticity of the lower extremities (Ashworth score 3 or 4), having an acute MS attack or a history of an attack in the last 1 month, having an orthopedic or systemic problem that would prevent participation in the tests, having another neuromuscular disorder other than MS, visual involvement or diplopia, and is that he has a cardio-pulmonary problem that will prevent him from participating in the tests.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals who applied to Fırat University Training and Research Hospital and were diagnosed with Relapsin-Remitting MS by a neurologist will be included in our study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-04-18 (Estimated); Study Completion 2022-05-09 (Estimated)

PRIMARY OUTCOMES:
L test | 1 week
  It is an expanded version of the TUG and is designed to assess advanced functional ambulation with more detail available elsewhere. It is recorded when the participant gets up from the chair, walks 3 m to a cone, turns 90° to the right, continues to walk 7 m to the next cone, turns 180° left around the cone, then returns to the chair the same way. The test time is recorded, starting with the word "go" and ending with the participant's back touching the back of the chair.
Timed Get Up and Go Test | 1 week
  It is applied to assess the balance and fall risk of individuals. The patient is first asked to sit leaning on the chair. The patient is then asked to stand up, walk with regular steps for a predetermined distance of 3 meters, return at the end of 3 meters and sit in a chair. During the test, the patient's walking time is recorded in seconds with a stopwatch. The test was repeated three times and the average value will be recorded

SECONDARY OUTCOMES:
3-meter Walk Back Test | 1 week
  The 3-meter distance is marked with a black tape and participants are asked to align their heels with the black tape. Individuals are asked to walk backwards as soon as possible with the "walk" command and stop when they reach 3 meters. Meanwhile, the elapsed time is recorded in seconds. Evaluation will be done three times and average time will be recorded
10-Meter Walk Test (10MeWT) | 1 week
  The 10MeWT was measured concurrently in the 2MWT (10MeWT-2M) and 6MWT (10MeWT-6M) to obtain the walking speeds of the participants. One reason for the simultaneous measurements was that the test protocols and the environmental set-up of the 2MWT, 6MWT and 10MeWT were very similar. Combining these tests could reduce the number of repeated walking and the resulting fatigue for the participants, and thus maximized their compliance to the tests. The walking speeds achieved in the 2MWT (10MeWT-2M) and 6MWT (10MeWT-6M) were treated as distinctive outcomes and analyzed separately because we believed that the instructions given to the participants in the 2MWT and 6MWT were different, possibly resulting in differences in the timed walk tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat university, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frohman EM, Racke MK, Raine CS. Multiple sclerosis--the plaque and its pathogenesis. N Engl J Med. 2006 Mar 2;354(9):942-55. doi: 10.1056/NEJMra052130. No abstract available. PMID 16510748
- [Background] Frzovic D, Morris ME, Vowels L. Clinical tests of standing balance: performance of persons with multiple sclerosis. Arch Phys Med Rehabil. 2000 Feb;81(2):215-21. doi: 10.1016/s0003-9993(00)90144-8. PMID 10668778
- [Background] Williams NP, Roland PS, Yellin W. Vestibular evaluation in patients with early multiple sclerosis. Am J Otol. 1997 Jan;18(1):93-100. PMID 8989958
- [Background] Daley ML, Swank RL. Quantitative posturography: use in multiple sclerosis. IEEE Trans Biomed Eng. 1981 Sep;28(9):668-71. doi: 10.1109/TBME.1981.324761. No abstract available. PMID 7319527
- [Background] Lanzetta D, Cattaneo D, Pellegatta D, Cardini R. Trunk control in unstable sitting posture during functional activities in healthy subjects and patients with multiple sclerosis. Arch Phys Med Rehabil. 2004 Feb;85(2):279-83. doi: 10.1016/j.apmr.2003.05.004. PMID 14966714
- [Background] Cattaneo D, De Nuzzo C, Fascia T, Macalli M, Pisoni I, Cardini R. Risks of falls in subjects with multiple sclerosis. Arch Phys Med Rehabil. 2002 Jun;83(6):864-7. doi: 10.1053/apmr.2002.32825. PMID 12048669
- [Background] Guideline for the prevention of falls in older persons. American Geriatrics Society, British Geriatrics Society, and American Academy of Orthopaedic Surgeons Panel on Falls Prevention. J Am Geriatr Soc. 2001 May;49(5):664-72. No abstract available. PMID 11380764
- [Background] DeBolt LS, McCubbin JA. The effects of home-based resistance exercise on balance, power, and mobility in adults with multiple sclerosis. Arch Phys Med Rehabil. 2004 Feb;85(2):290-7. doi: 10.1016/j.apmr.2003.06.003. PMID 14966716
- [Background] Cattaneo D, Cardini R. Computerized system to improve voluntary control of balance in neurological patients. Cyberpsychol Behav. 2001 Dec;4(6):687-94. doi: 10.1089/109493101753376632. PMID 11800176
- [Background] Cattaneo D, Marazzini F, Crippa A, Cardini R. Do static or dynamic AFOs improve balance? Clin Rehabil. 2002 Dec;16(8):894-9. doi: 10.1191/0269215502cr547oa. PMID 12501952
- [Background] Hobart JC, Riazi A, Lamping DL, Fitzpatrick R, Thompson AJ. Measuring the impact of MS on walking ability: the 12-Item MS Walking Scale (MSWS-12). Neurology. 2003 Jan 14;60(1):31-6. doi: 10.1212/wnl.60.1.31. PMID 12525714
- [Background] Tesio L, Perucca L, Franchignoni FP, Battaglia MA. A short measure of balance in multiple sclerosis: validation through Rasch analysis. Funct Neurol. 1997 Sep-Oct;12(5):255-65. PMID 9439943
- [Background] Smith PS, Hembree JA, Thompson ME. Berg Balance Scale and Functional Reach: determining the best clinical tool for individuals post acute stroke. Clin Rehabil. 2004 Nov;18(7):811-8. doi: 10.1191/0269215504cr817oa. PMID 15573838
- [Background] Tsang CS, Liao LR, Chung RC, Pang MY. Psychometric properties of the Mini-Balance Evaluation Systems Test (Mini-BESTest) in community-dwelling individuals with chronic stroke. Phys Ther. 2013 Aug;93(8):1102-15. doi: 10.2522/ptj.20120454. Epub 2013 Apr 4. PMID 23559522
- [Background] Breisinger TP, Skidmore ER, Niyonkuru C, Terhorst L, Campbell GB. The Stroke Assessment of Fall Risk (SAFR): predictive validity in inpatient stroke rehabilitation. Clin Rehabil. 2014 Dec;28(12):1218-24. doi: 10.1177/0269215514534276. Epub 2014 May 21. PMID 24849795
- [Background] Sebastiao E, Sandroff BM, Learmonth YC, Motl RW. Validity of the Timed Up and Go Test as a Measure of Functional Mobility in Persons With Multiple Sclerosis. Arch Phys Med Rehabil. 2016 Jul;97(7):1072-7. doi: 10.1016/j.apmr.2015.12.031. Epub 2016 Mar 2. PMID 26944709
- [Background] Nilsagard Y, Lundholm C, Gunnarsson LG, Dcnison E. Clinical relevance using timed walk tests and 'timed up and go' testing in persons with multiple sclerosis. Physiother Res Int. 2007 Jun;12(2):105-14. doi: 10.1002/pri.358. PMID 17536648
- [Background] Nguyen VC, Miller WC, Asano M, Wong RY. Measurement properties of the L test for gait in hospitalized elderly. Am J Phys Med Rehabil. 2007 Jun;86(6):463-8. doi: 10.1097/PHM.0b013e31805b8193. PMID 17515685
- [Background] Deathe AB, Miller WC. The L test of functional mobility: measurement properties of a modified version of the timed "up & go" test designed for people with lower-limb amputations. Phys Ther. 2005 Jul;85(7):626-35. PMID 15982169
- [Background] Kim JS, Chu DY, Jeon HS. Reliability and validity of the L test in participants with chronic stroke. Physiotherapy. 2015 Jun;101(2):161-5. doi: 10.1016/j.physio.2014.09.003. Epub 2014 Oct 28. PMID 25555897
- [Background] Lexell JE, Downham DY. How to assess the reliability of measurements in rehabilitation. Am J Phys Med Rehabil. 2005 Sep;84(9):719-23. doi: 10.1097/01.phm.0000176452.17771.20. PMID 16141752
- [Background] Haas B, Clarke E, Elver L, Gowman E, Mortimer E, Byrd E. The reliability and validity of the L-test in people with Parkinson's disease. Physiotherapy. 2019 Mar;105(1):84-89. doi: 10.1016/j.physio.2017.11.218. Epub 2017 Dec 5. PMID 29395266
- [Background] Bilek F, Demir CF. Validity and reliability of the 3-meter backward walk test in mildly disabled persons with multiple sclerosis. Mult Scler Relat Disord. 2022 Feb;58:103532. doi: 10.1016/j.msard.2022.103532. Epub 2022 Jan 19. PMID 35066275
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Roos MA, Reisman DS, Hicks G, Rose W, Rudolph KS. Development of the Modified Four Square Step Test and its reliability and validity in people with stroke. J Rehabil Res Dev. 2016;53(3):403-12. doi: 10.1682/JRRD.2014.04.0112. PMID 27271003